CLINICAL TRIAL: NCT02417064
Title: A Randomized, Double-blind, Multicenter, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Fixed Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Subjects With Treatment-resistant Depression
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Fixed Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Participants With Treatment-resistant Depression
Acronym: TRANSFORM-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107146; ESKETINTRD3001 (Other: Janssen Research & Development, LLC); 2014-004584-20 (EudraCT Number)
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Treatment-resistant Depression
Keywords: Treatment-resistant Depression; Esketamine; Placebo; Oral Antidepressant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Duloxetine Hydrochloride; Antidepressive Agents; Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Intranasal Esketamine 84mg plus Oral Antidepressant (Experimental): As part of an initial titration, participants will self-administer 56 milligrams (mg) of esketamine intranasally on Day 1, and then 84 mg from Day 4 onwards, twice per week for 4 weeks as a fixed dose regimen in Double-Blind Induction Phase. In addition participants will simultaneously initiate a new, open-label oral antidepressant (i.e, duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Esketamine; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)
- Esketamine 56 mg plus Oral Antidepressant (Experimental): Starting from Day 1, participants will self-administer 56 mg of esketamine, intranasally, twice per week for 4 weeks as a fixed dose regimen in Double-Blind Induction Phase. In addition participants will simultaneously initiate a new, open-label oral antidepressant (i.e, duloxetine, escitalopram, sertraline, or venlafaxine XR) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Esketamine; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)
- Placebo plus Oral Antidepressant (Active Comparator): Participants will self-administer matching placebo, intranasally, twice per week for 4 weeks as a fixed dose regimen in Double-Blind Induction Phase. In addition participants will simultaneously initiate a new, open-label oral antidepressant (i.e, duloxetine, escitalopram, sertraline, or venlafaxine XR) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Placebo; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)

INTERVENTIONS:
Drug: Esketamine — Participants will self-administer either 84 mg or 56 mg of esketamine, intranasally, twice per week for 4 weeks as a fixed dose regimen in Double-Blind Induction Phase.
  Arms: Esketamine 56 mg plus Oral Antidepressant; Intranasal Esketamine 84mg plus Oral Antidepressant
Drug: Placebo — Participants will self-administer matching placebo, intranasally, twice per week for 4 weeks as a fixed dose regimen in Double-Blind Induction Phase.
  Arms: Placebo plus Oral Antidepressant
Drug: Duloxetine (Oral Antidepressant) — Duloxetine could be selected as the oral antidepressant medication by the investigator based on review of Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and relevant prior antidepressant medication information. The minimum therapeutic dose is 60 milligram per day (mg/day).
Drug: Escitalopram (Oral antidepressant) — Escitalopram could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Escitalopram will be titrated up to a dose of 20 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 10 mg/day.
Drug: Sertraline (Oral Antidepressant) — Sertraline could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Sertraline will be titrated up to a dose of 200 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 50 mg/day.
Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant) — Venlafaxine Extended Release could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Venlafaxine Extended Release will be titrated up to a dose of 225 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 150 mg/day.

SUMMARY:
The purpose of this study is to compare the efficacy and safety of switching treatment-resistant depression (TRD) participants from a prior antidepressant treatment (to which they have not responded) to either intranasal esketamine plus a new oral antidepressant or switching to a new oral antidepressant plus intranasal placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither the researchers nor the participants know what treatment the participant is receiving), active-controlled, multicenter study (more than 1 study site) in participants with TRD to assess the efficacy, safety, and tolerability of fixed doses of intranasal esketamine plus a newly initiated oral antidepressant compared with a newly initiated oral antidepressant (active comparator) plus intranasal placebo. The study will consist of 3 phases: Screening/Prospective Observational Phase (4-7 weeks), Double-blind Induction Phase (4-weeks), Follow-up Phase (24-weeks). Participants who rollover into a long-term maintenance study will not participate in the Follow-up Phase. At the start of the screening/prospective observational phase, the participant must have had documented non-response to at least 1 antidepressant treatment (based on Massachusetts General Hospital - Antidepressant Treatment Response Questionnair [MGH-ATRQ]) in the current episode of depression, and participant is taking a different oral antidepressant treatment on the MGH-ATRQ for at least the previous 2 weeks at or above the minimum therapeutic dose. This antidepressant treatment, as well as any other ongoing medications being taken for depression at screening (including adjunctive/ augmentation therapies), will continue from the start of Week 1 through the end of Week 4 of the screening/prospective observational phase. Participants will be randomly assigned to receive Intranasal esketamine (56 milligrams [mg]), Intranasal esketamine (84 mg), or Intranasal placebo. In addition, each participant will be assigned to receive 1 of 4 oral antidepressant medications from 2 different classes of antidepressant treatments, a Selective Serotonin Reuptake Inhibitor (SSRI) (escitalopram or sertraline) or a Serotonin and Norepinephrine Reuptake Inhibitor (SNRI) (duloxetine or venlafaxine extended release [XR]), initiated on Day 1 and continued through the double-blind induction phase. Participants will be primarily evaluated for improvement in depressive symptoms as assessed by change in Montgomery-Asberg Depression Rating Scale (MADRS) total score at Week 4. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form (ICF), participant must be a man or woman 18 (or older if the minimum legal age of consent in the country in which the study is taking place is greater than [>]18) to 64 years of age, inclusive
* At the start of the screening/prospective observational phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) (if single-episode MDD, the duration must be greater than or equal to [>=] 2 years) or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* At the start of the screening/prospective observational phase, participant must have an Inventory of Depressive Symptomatology-Clinician rated ( IDS-C30) total score of greater than or equal to (>=) 34
* At the start of the screening/prospective observational phase, participants must have had non-response (less than or equal to [<=25] percent [%] improvement) to >=1 but less than or equal to (<=) 5 (if current episode is >2 years, upper limit is applicable to only the last 2 years) oral antidepressant treatments taken at adequate dosage and for adequate duration, as assessed using the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and documented by medical history and pharmacy/prescription records, for the current episode of depression.

Participant is taking a different oral antidepressant treatment on the MGH-ATRQ for at least the previous 2 weeks at or above the minimum therapeutic dose

- The participant's current major depressive episode, depression symptom severity (Week 1 MADRS total score >=28 required), and antidepressant treatment response in the current depressive episode, must be confirmed using a Site Independent Qualification Assessment

Exclusion Criteria:

* Participants who have previously demonstrated nonresponse of depressive symptoms to esketamine or ketamine in the current major depressive episode, to all 4 of the oral antidepressant treatment options available for the double-blind induction phase (i.e, duloxetine, escitalopram, sertraline, and venlafaxine extended release [XR]) in the current major depressive episode (based on MGH-ATRQ), or an adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT
* Participant has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features bipolar or related disorders (confirmed by the MINI), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening/prospective observational phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Participants with history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (90):
- United States (37):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Garden Grove, California
  - Orange, California
  - San Diego, California
  - San Marcos, California
  - San Rafael, California
  - Bradenton, Florida
  - Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Maywood, Illinois
  - Schaumburg, Illinois
  - Wichita, Kansas
  - Gaithersburg, Maryland
  - Boston, Massachusetts
  - Quincy, Massachusetts
  - Watertown, Massachusetts
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - O'Fallon, Missouri
  - Saint Charles, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Lincoln, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Woodstock, Vermont
  - Bothell, Washington
  - Middleton, Wisconsin
- Belgium (9):
  - Aalst
  - Bruges
  - Brussels
  - Ghent
  - Hasselt
  - Heusden-Zolder
  - Liège
  - Spa
  - Yvoir
- Brazil (7):
  - Belo Horizonte
  - Curitiba
  - Fortaleza
  - Passo Fundo
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
- Canada (6):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Estonia (3):
  - Pärnu
  - Tallinn
  - Tartu
- France (15):
  - Besançon
  - Clermont-Ferrand
  - Douai
  - Issy-les-Moulineaux
  - La Tronche
  - Lille
  - Limoges
  - Montpellier
  - Nantes
  - Neuilly-sur-Marne
  - Nîmes
  - Paris
  - Poitiers
  - Toulon
  - Tours
- Hungary (2):
  - Budapest
  - Vác
- Mexico (6):
  - Guadalajara
  - León
  - Mazatlán
  - Mexico City
  - Monterrey
  - San Luis Potosí City
- Slovakia (5):
  - Bratislava
  - Liptovský Mikuláš
  - Rimavská Sobota
  - Rožňava
  - Svidník

REFERENCES:
- [Derived] Kern Sliwa J, Naranjo RR Jr, Turkoz I, Petrillo MP, Cabrera P, Trivedi M. Effects of esketamine nasal spray on depressive symptom severity in adults with treatment-resistant depression and associations between the Montgomery-Asberg Depression Rating Scale and the 9-item Patient Health Questionnaire. CNS Spectr. 2024 Jun;29(3):176-186. doi: 10.1017/S1092852924000105. Epub 2024 Apr 1. PMID 38557430
- [Derived] Turkoz I, Nelson JC, Wilkinson ST, Borentain S, Macaluso M, Trivedi MH, Williamson D, Sheehan JJ, Salvadore G, Singh J, Daly E. Predictors of response and remission in patients with treatment-resistant depression: A post hoc pooled analysis of two acute trials of esketamine nasal spray. Psychiatry Res. 2023 May;323:115165. doi: 10.1016/j.psychres.2023.115165. Epub 2023 Mar 16. PMID 37019044
- [Derived] Jha MK, Williamson DJ, Magharehabed G, Turkoz I, Daly EJ, Trivedi MH. Intranasal esketamine effectively treats treatment-resistant depression in adults regardless of baseline irritability. J Affect Disord. 2023 Jan 15;321:153-160. doi: 10.1016/j.jad.2022.10.020. Epub 2022 Oct 20. PMID 36273682
- [Derived] Chen G, Chen L, Zhang Y, Li X, Lane R, Lim P, Daly EJ, Furey ML, Fedgchin M, Popova V, Singh JB, Drevets WC. Relationship Between Dissociation and Antidepressant Effects of Esketamine Nasal Spray in Patients With Treatment-Resistant Depression. Int J Neuropsychopharmacol. 2022 Apr 19;25(4):269-279. doi: 10.1093/ijnp/pyab084. PMID 35022754
- [Derived] Jones RR, Freeman MP, Kornstein SG, Cooper K, Daly EJ, Canuso CM, Nicholson S. Efficacy and safety of esketamine nasal spray by sex in patients with treatment-resistant depression: findings from short-term randomized, controlled trials. Arch Womens Ment Health. 2022 Apr;25(2):313-326. doi: 10.1007/s00737-021-01185-6. Epub 2022 Jan 1. PMID 34973081
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Turkoz I, Daly E, Singh J, Lin X, Tymofyeyev Y, Williamson D, Salvadore G, Nash AI, Macaluso M, Wilkinson ST, Nelson JC. Treatment Response With Esketamine Nasal Spray Plus an Oral Antidepressant in Patients With Treatment-Resistant Depression Without Evidence of Early Response: A Pooled Post Hoc Analysis of the TRANSFORM Studies. J Clin Psychiatry. 2021 Jul 20;82(4):20m13800. doi: 10.4088/JCP.20m13800. PMID 34288609
- [Derived] Doty RL, Popova V, Wylie C, Fedgchin M, Daly E, Janik A, Ochs-Ross R, Lane R, Lim P, Cooper K, Melkote R, Jamieson C, Singh J, Drevets WC. Effect of Esketamine Nasal Spray on Olfactory Function and Nasal Tolerability in Patients with Treatment-Resistant Depression: Results from Four Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Studies. CNS Drugs. 2021 Jul;35(7):781-794. doi: 10.1007/s40263-021-00826-9. Epub 2021 Jul 7. PMID 34235612
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208
- [Derived] Katz EG, Hough D, Doherty T, Lane R, Singh J, Levitan B. Benefit-Risk Assessment of Esketamine Nasal Spray vs. Placebo in Treatment-Resistant Depression. Clin Pharmacol Ther. 2021 Feb;109(2):536-546. doi: 10.1002/cpt.2024. Epub 2020 Oct 13. PMID 32860422
- [Derived] Saad Z, Hibar D, Fedgchin M, Popova V, Furey ML, Singh JB, Kolb H, Drevets WC, Chen G. Effects of Mu-Opiate Receptor Gene Polymorphism rs1799971 (A118G) on the Antidepressant and Dissociation Responses in Esketamine Nasal Spray Clinical Trials. Int J Neuropsychopharmacol. 2020 Dec 3;23(9):549-558. doi: 10.1093/ijnp/pyaa030. PMID 32367114
- [Derived] Fedgchin M, Trivedi M, Daly EJ, Melkote R, Lane R, Lim P, Vitagliano D, Blier P, Fava M, Liebowitz M, Ravindran A, Gaillard R, Ameele HVD, Preskorn S, Manji H, Hough D, Drevets WC, Singh JB. Efficacy and Safety of Fixed-Dose Esketamine Nasal Spray Combined With a New Oral Antidepressant in Treatment-Resistant Depression: Results of a Randomized, Double-Blind, Active-Controlled Study (TRANSFORM-1). Int J Neuropsychopharmacol. 2019 Oct 1;22(10):616-630. doi: 10.1093/ijnp/pyz039. PMID 31290965
- See also: A Randomized, Double-blind, Multicenter, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Fixed Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Subjects with Treatment-resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107146&attachmentIdentifier=0cb41e2c-8076-43c1-8eb1-ae4e9fe0b016&fileName=ESKETINTRD3001_(CR107146)_Additional_Results_Data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Esketamine 56 mg Plus Oral Antidepressant: Participants self-administered 56 milligram (mg) of intranasal esketamine (Esk) twice per week for 4 weeks in double-blind (DB) induction phase. Also, participants simultaneously initiated new oral antidepressant (AD) with one of following: duloxetine (60 mg/day- Weeks 1, 2, 3 and 4), escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2 to 4 with minimum therapeutic dose [MTD] of 10 mg/day), sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MTD of 50 mg/day) or venlafaxine extended release (XR) (75 mg/day- Week 1, 150 mg/day- Week 2, 225 mg/day- Weeks 3 and 4 with MTD of 150 mg/day) on Day 1 taken daily in DB induction phase. Participants who were not eligible or chose to not participate in maintenance of effect study (ESKETINTRD3003 [NCT02493868]) and had received at least 1 dose of intranasal Esk 56 mg+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks.
- Intranasal Esketamine 84 mg Plus Oral AD: Participants self-administered 56 mg of intranasal esketamine on Day 1 and then 84 mg from Day 4 onwards twice per week for 4 Weeks in DB induction phase. Also, participants simultaneously initiated new oral AD with one of following: duloxetine (60 mg/day- Weeks 1, 2, 3 and 4), escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2 to 4 with minimum therapeutic dose [MTD] of 10 mg/day), sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MTD of 50 mg/day) or venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, 225 mg/day- Weeks 3 and 4 with MTD of 150 mg/day) on Day 1 taken daily in DB induction phase. Participants who were not eligible or chose to not participate in maintenance of effect study (ESKETINTRD3003) and had received at least 1 dose of intranasal Esk 84 mg+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks.
- Oral AD Plus Intranasal Placebo: Participants self-administered intranasal matching placebo, twice per week for 4 weeks in DB induction phase. Also, participants simultaneously initiated new oral AD with one of following: duloxetine (60 mg/day- Weeks 1, 2, 3 and 4), escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2 to 4 with minimum therapeutic dose [MTD] of 10 mg/day), sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MTD of 50 mg/day) or venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, 225 mg/day- Weeks 3 and 4 with MTD of 150 mg/day) on Day 1 taken daily in DB induction phase. Participants who were not eligible or chose to not participate in maintenance of effect study (ESKETINTRD3003) and had received at least 1 dose of intranasal placebo+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks.
Period: Double-blind Induction Phase (4 Weeks)
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Started | 117 | 116 | 113
Full Analysis Set (FAS) | 115 | 114 | 113
Safety Analysis Set | 115 | 116 | 113
Completed | 111 | 97 | 107
Not Completed | 6 | 19 | 6
Not completed — Adverse Event | 1 | 7 | 2
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 1
Not completed — Other | 1 | 4 | 2
Period: Follow-up Phase (24 Weeks)
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Started | 47 | 52 | 69
Completed | 8 | 10 | 18
Not Completed | 39 | 42 | 51
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 9 | 2
Not completed — PI Decision | 34 | 29 | 44
Not completed — Other | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least 1 dose of intranasal study medication or
  1 dose of oral antidepressant medication during the double-blind induction phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo | Total
Number analyzed (Participants) | 115 | 116 | 113 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 115 | 115 | 112 | 342
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.18) | 45.7 (11.02) | 46.8 (11.36) | 46.3 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 80 | 81 | 242
  Male | 34 | 36 | 32 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 27 | 31 | 91
  Not Hispanic or Latino | 74 | 80 | 71 | 225
  Unknown or Not Reported | 8 | 9 | 11 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 2 | 5
  Black or African American | 7 | 8 | 5 | 20
  White | 91 | 86 | 86 | 263
  More than one race | 8 | 11 | 11 | 30
  Unknown or Not Reported | 7 | 9 | 9 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 8 | 9 | 12 | 29
  Brazil | 20 | 19 | 18 | 57
  Canada | 7 | 7 | 6 | 20
  Estonia | 3 | 4 | 3 | 10
  France | 11 | 10 | 10 | 31
  Hungary | 3 | 2 | 1 | 6
  Mexico | 14 | 16 | 15 | 45
  Slovakia | 4 | 3 | 3 | 10
  United States | 45 | 46 | 45 | 136

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score up to Day 28 of Double- Blind Induction Phase- Mixed- Effects Model Using Repeated Measures (MMRM) Analysis
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Baseline up to Day 28 of Double-blind Induction Phase
Population: Full analysis set (FAS): all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral antidepressant medication during double-blind induction phase. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 111 | 98 | 108
Units on a scale | -19.0 (13.86) | -18.8 (14.12) | -14.8 (15.07)
Statistical Analysis 1: Comparison: Intranasal Esketamine 84 mg Plus Oral AD vs Oral AD Plus Intranasal Placebo; Test type: Superiority; p = 0.088, Mixed Model for Repeated Measures; Difference of Least Square (LS) Means = -3.2, 95% CI 2-sided [-6.88 to 0.45]
Statistical Analysis 2: Comparison: Intranasal Esketamine 56 mg Plus Oral Antidepressant vs Oral AD Plus Intranasal Placebo; Test type: Superiority; Difference of Least Square (LS) Means = -4.1, 95% CI 2-sided [-7.67 to -0.49]

2. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Missing data was imputed using Last Observation Carried Forward (LOCF) method and last post baseline observation during double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 115 | 113 | 113
Units on a scale | -18.3 (14.21) | -17.4 (14.25) | -14.3 (15.00)
Statistical Analysis 1: Comparison: Intranasal Esketamine 84 mg Plus Oral AD vs Oral AD Plus Intranasal Placebo; Test type: Superiority; p = 0.250, ANCOVA; Difference of Least Square (LS) Means = -2.0, 95% CI 2-sided [-5.52 to 1.42]
Statistical Analysis 2: Comparison: Intranasal Esketamine 56 mg Plus Oral Antidepressant vs Oral AD Plus Intranasal Placebo; Test type: Superiority; Difference of Least Square (LS) Means = -4.1, 95% CI 2-sided [-7.53 to -0.6]

3. Secondary Outcome: Percentage of Participants With Onset of Clinical Response by Day 2 and Day 8
Description: A participant was defined as having a clinical response if there was at least 50% improvement (decrease) from baseline in the MADRS total score with onset by Day 2 and Day 8 that was maintained to Day 28. Participants were allowed one excursion (non-response) on Days 8, 15 or 22, however score must show at least 25% improvement. Participants who did not meet these criteria or discontinued during the study before Day 28 were considered as non-responders and were assigned the value of 0 (that is no). MADRS is clinician-rated scale that consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), for total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Day 2 up to Day 28 and Day 8 up to Day 28
Population: FAS: all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during the double-blind induction phase.
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 115 | 114 | 113
Percentage of Participants
  Day 2 up to Day 28 | 10.4 | 8.8 | 1.8
  Day 8 up to Day 28 | 13.0 | 11.4 | 3.5

4. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score up to Day 28 of Double-blind Induction Phase- MMRM Analysis
Description: The SDS is a participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. The first 3 items assess disruption of 1) work/school, 2) social life, and 3) family life/home responsibilities using 0 (not at all) to 10 (extremely) rating scale. Score for first 3 items are summed to create total score of 0 (unimpaired) to 30 (highly impaired), where higher score indicates greater impairment.
Time Frame: Baseline up to Day 28 of Double-blind Induction phase
Population: FAS: all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during the double-blind induction phase. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 88 | 87 | 90
Units on a scale | -11.0 (9.32) | -11.1 (10.04) | -8.4 (9.70)

5. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis
Description: The SDS is a participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. The first 3 items assess disruption of 1) work/school, 2) social life, and 3) family life/home responsibilities using 0 (not at all) to 10 (extremely) rating scale. Score for first 3 items are summed to create total score of 0 (unimpaired) to 30 (highly impaired) where higher score indicates greater impairment. Missing data was imputed using LOCF method and the last post baseline observation during the double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 91 | 99 | 95
Units on a scale | -10.7 (9.39) | -10.2 (10.00) | -8.1 (9.57)

6. Secondary Outcome: Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Total Score up to Day 28 of Double-blind Induction Phase- MMRM Analysis
Description: PHQ-9 is 9-item, self-reported scale assessing 9 symptom domains of Diagnostic and Statistical Manual of Mental Disorders, Major Depressive Disorder criteria. Each item is rated on 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half days, 3 = Nearly every day). The scores are summed for a total score ranging from 0-27. Higher score indicates greater severity of depression. Severity of PHQ-9 categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19), Severe (20-27). The recall period is 2 weeks.
Time Frame: Baseline up to Day 28 of Double-blind Induction phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 110 | 99 | 108
Units on a scale | -11.0 (8.07) | -11.7 (7.74) | -9.1 (8.35)

7. Secondary Outcome: Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis
Description: PHQ-9 is 9-item, self-reported scale assessing 9 symptom domains of Diagnostic and Statistical Manual of Mental Disorders, Major Depressive Disorder criteria. Each item is rated on 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half days, 3 = Nearly every day). The scores are summed for a total score ranging from 0-27. Higher score indicates greater severity of depression. Severity of PHQ-9 categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19), Severe (20-27). The recall period is 2 weeks. Missing data was imputed using LOCF method and the last post baseline observation during the double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 113 | 112 | 113
Units on a scale | -10.9 (8.26) | -10.9 (7.81) | -8.9 (8.37)

8. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Reduction From Baseline in MADRS Total Score at Day 28 of Double-blind Induction Phase (Observed Data)
Description: A participant was defined as a responder (yes=1 and no=0) at a given time point if the percent reduction from baseline in MADRS total score is at least 50 percent (%). The percentage of participants who achieved at least 50% reduction from baseline were reported. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: At Day 28 of Double-blind Induction phase
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 111 | 98 | 108
Percentage of Participants | 54.1 | 53.1 | 38.9

9. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Reduction From Baseline in MADRS Total Score at the Endpoint (Double-blind Induction Phase [Day 28]) (LOCF Data)
Description: A participant was defined as a responder (yes=1 and no=0) at a given time point if the percent reduction from baseline in MADRS total score is at least 50 percent (%). The percentage of participants who achieved at least 50% reduction from baseline were reported. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Missing data was imputed using LOCF method and the last post baseline observation during the double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: At Day 28 (Double-blind Endpoint)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 115 | 113 | 113
Percentage of Participants | 53.0 | 47.8 | 37.2

10. Secondary Outcome: Percentage of Participants in Remission (MADRS<=12) at Day 28 of Double-blind Induction Phase (Observed Data)
Description: Participants who had a MADRS total score of less than or equal to (<=) 12 were considered as remitters. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: At Day 28 of Double-blind Induction Phase
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 111 | 98 | 108
Percentage of participants | 36 | 38.8 | 30.6

11. Secondary Outcome: Percentage of Participants in Remission (MADRS<=12) at the Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis (LOCF Data)
Description: Participants who had a MADRS total score of less than or equal to (<=) 12 were considered as remitters. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Missing data was imputed using LOCF method and the last post baseline observation during the double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: At Day 28 (Double-blind Endpoint)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 115 | 113 | 113
Percentage of participants | 34.8 | 35.4 | 29.2

12. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score up to Endpoint (Double-blind Induction Phase [Day 28])
Description: CGI-S provides measure of severity of participant's illness including participant's history, psychosocial circumstances, symptoms, behavior and impact of symptoms on ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Considering total clinical experience, participant is assessed on severity of mental illness according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill patients (a decrease in score indicates improvement). Missing data was imputed using LOCF method and the last post baseline observation during the double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 4
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 115 | 113 | 113
Units on a scale | -2.0 [-5 to 1] | -2.0 [-5 to 1] | -1.0 [-6 to 3]

13. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder-7 Item (GAD-7) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])
Description: GAD-7 is a brief and validated 7-item self-reported assessment of overall anxiety. Participants responded to each item using a 4 point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15-21). Missing data was imputed using LOCF method and the last post baseline observation during the double-blind induction phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Double-blind Endpoint (Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 111 | 109 | 111
Units on a scale | -7.4 (5.94) | -7.7 (5.72) | -6.0 (6.01)

14. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) up to End of Double-blind Induction Phase (Day 28): Health Status Index
Description: EQ-5D-5L measures health outcome self-completed by respondents. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). The descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each has 5 levels (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses are used to generate Health Status Index (HSI). HSI range is -0.148 to 0.949, is anchored at 0 (dead) and 1 (full health).
Time Frame: Baseline up to End of Double-blind Induction Phase (Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 113 | 112 | 113
Units on a scale | 0.224 (0.2481) | 0.243 (0.2395) | 0.181 (0.2495)

15. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) up to End of Double-blind Induction Phase (Day 28): EQ-VAS
Description: EQ-5D-5L measures health outcome self-completed by respondents. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Time Frame: Baseline up to end of Double-blind induction phase (Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 113 | 112 | 113
Units on a scale | 20.9 (25.04) | 19.1 (26.86) | 14.9 (27.15)

16. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) up to End of Double-blind Induction Phase (Day 28): Sum Score
Description: EQ-5D-5L measures health outcome self-completed by respondents. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). The descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each has 5 levels (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses are used to generate Health Status Index (HSI). HSI range is -0.148 to 0.949, is anchored at 0 (dead) and 1 (full health). EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline up to end of Double-blind Induction phase (Day 28)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine 56 mg Plus Oral Antidepressant | Intranasal Esketamine 84 mg Plus Oral AD | Oral AD Plus Intranasal Placebo
Number analyzed (Participants) | 113 | 112 | 113
Units on a scale | -19.0 (18.84) | -19.4 (18.43) | -14.6 (19.78)

ADVERSE EVENTS:
Time Frame: Up to follow up phase (Week 24)
Description: The population analyzed included safety analysis set- all randomized participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant medication during double-blind induction phase and follow-up analysis set- all participants who entered the follow-up phase and were evaluated for the safety.
Groups:
- DB Phase: Intranasal Esk 56 mg + Oral AD: Participants self-administered 56 mg of intranasal esketamine (Esk) twice per week for 4 weeks in double-blind (DB) induction phase. Also, participants simultaneously initiated new oral antidepressant (AD) with one of following: duloxetine (60 [milligram] mg/day- Weeks 1, 2, 3 and 4), escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2 to 4 with minimum therapeutic dose [MTD] of 10 mg/day), sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MTD of 50 mg/day) or venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, 225 mg/day- Weeks 3 and 4 with MTD of 150 mg/day) on Day 1 taken daily in DB induction phase.
- DB Phase: Intranasal Esk 84 mg + Oral AD: Participants self-administered 56 mg of intranasal esketamine on Day 1 and then 84 mg from Day 4 onwards twice per week for 4 Weeks in DB induction phase. Also, participants simultaneously initiated new oral AD with one of following: duloxetine (60 mg/day- Weeks 1, 2, 3 and 4), escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2 to 4 with minimum therapeutic dose [MTD] of 10 mg/day), sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MTD of 50 mg/day) or venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, 225 mg/day- Weeks 3 and 4 with MTD of 150 mg/day) on Day 1 taken daily in DB induction phase.
- DB Phase: Oral AD + Intranasal Placebo: Participants self-administered intranasal matching placebo, intranasally, twice per week for 4 weeks in DB induction phase. Also, participants simultaneously initiated new oral AD with one of following: duloxetine (60 mg/day- Weeks 1, 2, 3 and 4), escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2 to 4 with minimum therapeutic dose [MTD] of 10 mg/day), sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MTD of 50 mg/day) or venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, 225 mg/day- Weeks 3 and 4 with MTD of 150 mg/day) on Day 1 taken daily in DB induction phase.
- FU Phase: Intranasal Esk 56 mg + Oral AD: Participants who were not eligible or chose to not participate in maintenance of effect study (ESKETINTRD3003) and had received at least 1 dose of intranasal Esk 56 mg+ Oral AD in DB induction phase were followed in posttreatment follow-up (FU) phase for up to 24 weeks to assess safety and tolerability including withdrawal symptoms of study drug and for collection of additional informative data to assess the course of the participant's major depressive episode over a 24-week period.
- FU Phase: Intranasal Esk 84 mg + Oral AD: Participants who were not eligible or chose to not participate in maintenance of effect study (ESKETINTRD3003) and had received at least 1 dose of intranasal Esk 84 mg+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks to assess safety and tolerability including withdrawal symptoms of study drug and for collection of additional informative data to assess the course of the participant's major depressive episode over a 24-week period.
- FU Phase: Oral AD + Intranasal Placebo: Participants who were not eligible or chose to not participate in maintenance of effect study (ESKETINTRD3003) and had received at least 1 dose of intranasal placebo+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks to assess safety and tolerability including withdrawal symptoms of study drug and for collection of additional informative data to assess the course of the participant's major depressive episode over a 24-week period.
Arm/Group | DB Phase: Intranasal Esk 56 mg + Oral AD | DB Phase: Intranasal Esk 84 mg + Oral AD | DB Phase: Oral AD + Intranasal Placebo | FU Phase: Intranasal Esk 56 mg + Oral AD | FU Phase: Intranasal Esk 84 mg + Oral AD | FU Phase: Oral AD + Intranasal Placebo
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/116 | 0/113 | 0/47 | 0/52 | 0/69
Serious Adverse Events (participants affected / at risk) | 2/115 | 0/116 | 0/113 | 2/47 | 2/52 | 1/69
Other Adverse Events (participants affected / at risk) | 93/115 | 92/116 | 64/113 | 7/47 | 4/52 | 7/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Intranasal Esk 56 mg + Oral AD (N=115) | DB Phase: Intranasal Esk 84 mg + Oral AD (N=116) | DB Phase: Oral AD + Intranasal Placebo (N=113) | FU Phase: Intranasal Esk 56 mg + Oral AD (N=47) | FU Phase: Intranasal Esk 84 mg + Oral AD (N=52) | FU Phase: Oral AD + Intranasal Placebo (N=69)
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Intranasal Esk 56 mg + Oral AD (N=115) | DB Phase: Intranasal Esk 84 mg + Oral AD (N=116) | DB Phase: Oral AD + Intranasal Placebo (N=113) | FU Phase: Intranasal Esk 56 mg + Oral AD (N=47) | FU Phase: Intranasal Esk 84 mg + Oral AD (N=52) | FU Phase: Oral AD + Intranasal Placebo (N=69)
Vertigo (Ear and labyrinth disorders) | 24 | 24 | 2 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 8 | 9 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 3 | 0 | 1 | 2
Hypoaesthesia Oral (Gastrointestinal disorders) | 16 | 12 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 31 | 37 | 12 | 2 | 1 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 9 | 1 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 14 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 12 | 8 | 5 | 0 | 0 | 1
Feeling Drunk (General disorders) | 7 | 3 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 8 | 11 | 5 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 32 | 26 | 10 | 0 | 1 | 1
Dizziness Postural (Nervous system disorders) | 7 | 7 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 17 | 20 | 17 | 0 | 0 | 0
Headache (Nervous system disorders) | 23 | 24 | 19 | 4 | 2 | 3
Hypoaesthesia (Nervous system disorders) | 14 | 16 | 2 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 7 | 5 | 1 | 0 | 0 | 0
Mental Impairment (Nervous system disorders) | 6 | 3 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 19 | 11 | 3 | 0 | 0 | 0
Sedation (Nervous system disorders) | 6 | 8 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 24 | 21 | 13 | 0 | 0 | 0
Tremor (Nervous system disorders) | 4 | 6 | 2 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 10 | 9 | 7 | 1 | 0 | 2
Dissociation (Psychiatric disorders) | 30 | 32 | 4 | 0 | 0 | 0
Euphoric Mood (Psychiatric disorders) | 8 | 2 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 10 | 8 | 11 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 6 | 2 | 1 | 0 | 0 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 7 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 4 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Transient, dissociative effects of esketamine are difficult to blind, site staff who observed treatment sessions could have been biased. To ensure unbiased efficacy evaluations, independent, remote, blinded MADRS raters assessed treatment response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT02417064/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02417064/SAP_001.pdf